CLINICAL TRIAL: NCT00602797
Title: Phase II Study of Weekly Vinorelbine and Paclitaxel in Elderly Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Vinorelbine Tartrate and Paclitaxel in Treating Older Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0339-07-FB; NCI-2009-01584 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Taxes; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vinorelbine tartrate, paclitaxel) (Experimental): Patients receive vinorelbine tartrate IV over 6-10 minutes and paclitaxel IV over 1 hour once weekly for 6 weeks.
  Interventions: Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vinorelbine Tartrate

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Vinorelbine Tartrate — Given IV
  Other Names: Biovelbin; Eunades; KW-2307; Navelbine; Navelbine Ditartrate; Vinorelbine Ditartrate

SUMMARY:
This phase II trial studies the side effects and how well vinorelbine tartrate and paclitaxel works in treating older patients with non-small cell lung cancer that has spread to other placed in the body. Drugs used in chemotherapy, such as vinorelbine tartrate and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To assess the safety and efficacy of a combination of vinorelbine and paclitaxel administered weekly to elderly patients with advanced non-small cell lung cancer. II. To assess the response rate of a combination of vinorelbine and paclitaxel administered weekly to elderly patients with advanced non-small cell lung cancer. III. To assess the quality of life of elderly patients with advanced non-small cell lung cancer during administration of weekly paclitaxel and vinorelbine. OUTLINE: Patients receive vinorelbine tartrate intravenously (IV) over 6-10 minutes and paclitaxel IV over 1 hour once weekly for 6 weeks. Treatment repeats every 8 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven non-small cell lung cancer with evidence of distant metastases/malignant pleural effusion
* Measurable disease on imaging studies in 2 dimensions
* No previous therapy with either paclitaxel or vinorelbine, or any chemotherapy for the past five years
* Patients who have had a previous resection for their lung cancer and present with recurrent disease will be eligible
* Patients with other prior malignancies will be included, provided they have been disease-free for at least five years
* Patients with adequately treated basal cell or squamous cell carcinoma of the skin, adequately treated carcinoma in-situ of the cervix and hormone sensitive prostate cancer will be eligible
* Karnofsky score >= 70 (Eastern Cooperative Oncology Group [ECOG] 0-2)
* White blood cell (WBC) count >= 3,500/mm^3, OR
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelet count >= 100,000/mm^3
* Serum creatinine less than 1.5 times the upper limits of normal
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 1.5 times the upper limits of normal
* Serum alkaline phosphatase less than 2.5 times the upper limits of normal
* No active serious infections or other condition precluding chemotherapy
* Non-pregnant and non-nursing
* Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on the study
* Able to give informed consent
* Able to return for treatment and follow-up as specified in the protocol

Exclusion Criteria:

* Known hypersensitivity to any component of vinorelbine or paclitaxel or other required drugs in the study
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Inability to fulfill the requirements of the protocol

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apar K Ganti, MD, Principal Investigator — University of Nebraska
Locations (5):
- United States (5):
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Veterans Administration Medical Center, Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Huerter MM, Meza JL, Copur MS, Tolentino A, Marr AS, Ketcham M, DeSpiegelaere H, Kruse S, Kos ME, Swenson K, Radniecki SE, Kessinger A, Ganti AK. Weekly vinorelbine and paclitaxel in older patients with advanced non-small cell lung cancer: A phase II Fred and Pamela Buffet Cancer Center Clinical Trials Network study. J Geriatr Oncol. 2017 Jan;8(1):18-22. doi: 10.1016/j.jgo.2016.07.006. Epub 2016 Aug 1. PMID 27491498

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: This is a non-randomized, single-arm, phase II study of vinorelbine and paclitaxel in older patients with advanced non-small cell lung cancer. Vinorelbine (22.5 mg/m2) and paclitaxel (40 mg/m2) were given weekly for six weeks followed by a two-week break. Each patient received a maximum of two cycles (12 doses) of chemotherapy. All patients received standard premedication for nausea and hypersensitivity prophylaxis per individual institutional guidelines. Quality of life (QoL) was assessed at baseline, week 9, and week 17 using the Functional Assessment of Cancer Therapy lung cancer subscale instrument (FACT-L).
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vinorelbine Tartrate, Paclitaxel)
Number analyzed (Participants) | 20
Age, Customized [Mean (Standard Deviation); unit: years] — Age in years. Patients >70 years were eligible
  years | 76.9 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival.
Description: Time from first therapy until first documentation of clinical progression, relapse or death. Progression was defined as per RECIST v1.0 criteria as an at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions. The Kaplan-Meier method will be used to estimate time to event distributions.
Time Frame: Time from first therapy until first documentation of clinical progression, relapse or death assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment Group: Patients >70 years with advanced NSCLC treated with weekly paclitaxel and vinorelbine
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Months | 7.8 [1.92 to 13.56]

2. Secondary Outcome: Incidence of >Grade 3 Treatment-Emergent Non-hematological Adverse Events
Description: Toxicity will be assessed at the 0.05 two-sided level of significance. The Common Terminology Criteria for Adverse Events Version 3.0 will be used to grade the severity of adverse events.
Time Frame: Up to week 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
Participants | 6
Statistical Analysis 1: Comparison: Treatment; Adverse events will be graded using the NCI Common Toxicity Criteria (version 3.0); Test type: Other — An interim analysis was conducted after 10 patients were accrued. Since response rate seen at the first interim analysis was superior to that seen with standard of care, a new monitoring rule was approved. Toxicity monitoring would occur after 19 patients. If 6/19 patients had ≥grade 4 non-hematological toxicity, accrual will be terminated. This will provide 84% power to detect 40% toxicity; Proportion = 6 — If 6/19 patients had ≥grade 4 non-hematological toxicity, accrual will be terminated

3. Secondary Outcome: Response Rate Based on RECIST Criteria
Description: The measurement of effect will be based on the Response Evaluation Criteria In Solid Tumors criteria. Response rate is the sum of complete and partial responses. Complete Response is defined as the disappearance of all target lesions. Partial Response is defined as an at least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants | 5

ADVERSE EVENTS:
Description: All cause mortality is reported for the 20 patients enrolled in the study. Adverse event and Serious adverse events reporting is out of the 19 patients that were treated on the study. One of the patients enrolled on this study deteriorated before treatment and was not treated on the study.
Arm/Group | Treatment (Vinorelbine Tartrate, Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 16/20
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vinorelbine Tartrate, Paclitaxel) (N=19)
Febrile neutropenia (Infections and infestations) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Ischemic encephalopathy (Nervous system disorders) | 1 (1)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Vinorelbine Tartrate, Paclitaxel) (N=19)
Anemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 1
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 5
Febrile neutropenia (Infections and infestations) | 1
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 5
back pain (Musculoskeletal and connective tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
weakness (General disorders) | 1
fatigue (General disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Bowel perforation (Gastrointestinal disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Weight loss (Metabolism and nutrition disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Allergic reaction (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No